CLINICAL TRIAL: NCT02916797
Title: Effects of Stepping Training With and Without the Use of Visually Weight-taking Machine (VWTM) on Walking and Balance Ability in Patients With Stroke
Brief Title: Stepping Training Using Feedback in Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Khon Kaen University (Other)
Responsible Party: Principal Investigator, Sugalya Amatachaya, Assoc. Prof. Dr., Khon Kaen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PHD56I0044
Record Dates: First submitted 2016-09-22; First posted 2016-09-27 (Estimated); Last update posted 2019-03-12 (Actual); Status verified 2017-08

CONDITIONS: Cerebrovascular Accident
Keywords: Feedback; Physical Therapy
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Stepping training with feedback (Experimental): Subjects stand in a step standing position with placing the affected leg on the load cells of the VWTM and the non-affected leg slightly backward outside the load cells, look forward to light bars of the displayed section which will be set at their eye level. Then subjects will be instructed to shift/take their body-weight onto the affected leg until the green zone of the displayed section is lighting and a beep sound to alarm the subjects to step the non-affected leg forward and backward as much as they can. Subjects repetitively practice the task for 30 minutes with a period of sufficient rest as required.
  Interventions: Other: Stepping training with feedback
- Stepping training without feedback (No Intervention): Subjects will be trained and instructed the same as the experimental group but without using the displayed section, for approximately 30 minutes/day (excluding rest periods), 5 days/week, for 4 week. Then, every subject will be trained to walk overground with or without a walking device for 10 minutes in order to promote transferability of the part-task practice to the whole/target task. Subjects still receive routine treatments from other rehabilitation professionals as needed during participation in the study.

INTERVENTIONS:
Other: Stepping training with feedback — Stepping training with the use of external feedback. The subjects will be instructed to shift/take their body-weight onto the affected leg until the green zone of the displayed section is lighting and a beep sound to alarm the subjects to step the non-affected leg forward and backward as much as they can.
  Arms: Stepping training with feedback

SUMMARY:
* Are there differences in immediate effects of stepping training with and without the use of visually weight-taking machine (VWTM) on variables relating to well-controlled walking and walking symmetry in ambulatory patients with stroke?
* Are there differences of 4-week stepping training with and without the use of VWTM on variables relating to well-controlled walking and walking symmetry in ambulatory patients with stroke?

DETAILED DESCRIPTION:
* To compare immediate effects of stepping training with or without the use of VWTM on variables relating to well-controlled walking and walking symmetry in ambulatory patients with stroke.
* To compare effects of 4-week stepping training with or without the use of VWTM on variables relating to well-controlled walking and walking symmetry in patients with stroke.

ELIGIBILITY:
Inclusion Criteria:

* Subjects are independent ambulatory patients with first stroke episode with the age at least 45-74 years old,
* subacute (post-stroke time < 6 months) or chronic (post-stroke time ≥ 6 months) stroke
* Independent walking at least 10 meters with or without a walking device
* Able to follow verbal command used in this study

Exclusion Criteria:

* The subjects who have other medical conditions that might affect participation in the study such as uncontrolled underlying diseases (i.e. hypertension, heart disease, thyroid, etc.), deformity in the lower extremities, pain more than 5 out of 10 on a visual analog scale, legally blind or had a history of visual deficits that were unable to be corrected by glasses or contact lens, have a color blindness and inability to communicate or follow the commands used in this study

Ages: 45 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2016-04-10 (Actual); Primary Completion 2018-02-28 (Actual); Study Completion 2018-02-28 (Actual)

PRIMARY OUTCOMES:
10MWT | 4 weeks
  Walking speed

SECONDARY OUTCOMES:
6MWT | 4 weeks
  Walking endurance
TUGT | 4 weeks
  Balance and walking ability
Lower limb support ability | 4 weeks
  % of bosy-weight on single leg during stepping

CONTACTS AND LOCATIONS:
Overall Officials: Sugalya Amatachay, Ph.D., Principal Investigator — School of Physical Therapy,Faculty of Associated Medical Sciences, Khon Kaen University, Thailand

IPD SHARING:
Plan to Share IPD: No